CLINICAL TRIAL: NCT02868671
Title: Acupuncture Intervention in Subacute Mild Traumatic Brain Injury With Post-traumatic Stress Disorder: A Randomized Controlled Trial
Brief Title: Acupuncture for Mild Traumatic Brain Injury：A Functional Magnetic Resonance Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSFC81571752
Record Dates: First submitted 2016-07-21; First posted 2016-08-16 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2022-04

CONDITIONS: Acupuncture; Mild Traumatic Brain Injury; MRI
Keywords: mild TBI; post-concussion sydrome; Acupuncture
MeSH Terms: conditions — Brain Concussion | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- real acupuncture (Experimental): Participants will receive treatment four times a week for two weeks and three times a week for two weeks. Participants will be treated with major points: Yintang, Du20 (Bai Hui), LI4 (He Gu), LR3 (Tai Chong), ST36 (Zusanli) (front treatment) or GB20 (Feng Chi), SP6 (Sanyinjiao), BL15 (Xin Shu), BL18 (Gan Shu), BL23 (Shen Shu) (back treatment). The position of the treatment will alternate between sessions such that the first session will be on the back, with the next session on the front. In addition to the 5 required points, acupuncturist will be allowed to choose 1-3 more points. The supplemental points may be chosen from the following: HT7 (Shenmen), PC6 (Neiguan), SI3 (Hou Xi), RN6 (Qi Hai), KI 3 (Taixi), KI 6 (Zhao Hai), SP10 (Xue Hai), BL14 (Jue Yin Shu), BL17 (Ge Shu), BL20 (Pi Shu).
  Interventions: Other: acupuncture
- sham acupuncture (Sham Comparator): Participants randomized to sham acupuncture will receive a 'placebo' acupuncture session. For sham acupuncture, Streitberger needles, which acted like stage dagger with the shaft of the needle retracting into the handle, were placed at non-acupuncture points with the same number of acupuncture points in the VA group. The needle guiding tube will be used to create sensations that mimic needle manipulation.
  Interventions: Other: sham acupuncture
- No Intervention (No Intervention): All participants in this study will not receive interventions.

INTERVENTIONS:
Other: acupuncture
  Arms: real acupuncture
Other: sham acupuncture
  Arms: sham acupuncture

SUMMARY:
The overall goal of this study is to examine if acupuncture intervention can reduce the post-concussion symptom (PCS), and affective and cognitive complaints among mild traumatic brain injury (TBI). This study also hypothesized that compared to those in the sham acupuncture and waiting list control groups, patients in the real acupuncture group will have fewer symptoms of depression, sleep problems and post-concussion symptoms.

DETAILED DESCRIPTION:
Project Background: Acupuncture has been shown in other settings to alleviate symptoms of TBI that are reported to be precursors of post-concussion symptom, including affective (depression, anxiety) and somatic (headache, sleep difficulties) complaints. Evidence suggests that the increased intensity of these symptoms, particularly greater affective distress and injury-associated pain, increases vulnerability to neurodegenerative disease and PTSD. By treating post-TBI symptoms with acupuncture, these predisposing conditions will improve, and, as a result, the incidence of PCS in this patient population will be reduced.

Research plan: The overarching focus of this study is the use of acupuncture treatment, targeted to symptoms of mild TBI. The investigators propose a randomized, sham procedure and usual care-controlled clinical trial of acupuncture beginning at acute phase following mild traumatic brain injury (TBI). Participants meeting eligibility requirements will be randomized to 1 of 3 groups: verum acupuncture, sham acupuncture or waiting-list control. Acupuncture treatments will continue for one month, at which point all participants will be assessed for presence of mild TBI symptoms. Participants will be evaluated again after one-month acupuncture treatment and follow-up post-hospital discharge. The investigators hypothesize that true acupuncture will be more effective than sham acupuncture in reducing these outcomes at after treatment and follow-up stage. Patients were also scanned by 3T MRI scanner at baseline, one-month (after acupuncture treatment).

ELIGIBILITY:
Inclusion Criteria:

* subjects presenting to the study hospital emergency department (ED) after sustaining a acute head injury will be eligible if they:
* are aged 18-75 years;
* have a mild TBI, defined by the World Health Organization's Collaborating Centre for Neurotrauma Task Force (2005)
* no contraindications to MR
* injury within 7 days

Exclusion Criteria:

* experience with acupuncture treatment
* history of neurological disease, long-standing psychiatric condition, spinal cord injury, head injury, or a history of substance or alcohol abuse
* intubation and/or presence of a skull fracture
* administration of sedatives on arrival in the emergency department,
* the manifestation of mild traumatic brain injury (TBI) due to medications by other injuries (e.g., systemic injuries, facial injuries, or intubation) or other problems (e.g., psychological trauma, language barrier, or coexisting medical conditions), or caused by penetrating craniocerebral injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-08; Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Changes in PCS in patients following acupuncture treatments between baseline and after therapy | Baseline, after one-month therapy

SECONDARY OUTCOMES:
Changes in PCS in patients following acupuncture treatments between baseline and 6-12 months follow-up | Baseline, 6-12 months follow-up
Diffusion tensor magnetic metrics changes in patients following acupuncture treatment | baseline, one month

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes